CLINICAL TRIAL: NCT03172091
Title: Analysis of Volatile Organic Compounds in the Exhaled Air Breath of in Bilateral Lung Transplant Recipients Bi-pulmonary Transplant Patients: Search for Acute Rejection Markers
Brief Title: Volatile Organic Compounds as Markers of Acute Rejection in Lung Transplant
Acronym: VOC-TP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016/28; 2016-A00688-43 (Other: ANSM)
Record Dates: First submitted 2017-05-29; First posted 2017-06-01 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Transplant; Complication, Rejection
Keywords: Lung transplant; Acute resection; Volatile Organic Compounds
MeSH Terms: conditions — Rejection, Psychology | interventions — Electronic Nose; Spectrum Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute rejection (Experimental): Pulmonary transplant patients with acute rejection
  Interventions: Device: eNose (electronic nose); Device: Spectrometry
- Control group (Other): Pulmonary transplant patients without acute rejection
  Interventions: Device: eNose (electronic nose); Device: Spectrometry

INTERVENTIONS:
Device: eNose (electronic nose) — Collection of exhaled breath for an immediate analysis by electronic nose
Device: Spectrometry — Collection of exhaled breath for an immediate analysis by mass spectrometry

SUMMARY:
The aim of research is to identify markers of acute rejection by VOC analysis in exhaled breath of bilateral-lung transplanted patients. 120 bi-lung transplanted patients will be divided into two groups : patients with acute rejection diagnosed on transbronchial biopsies and patients with no acute rejection. Exhaled breath will be collected for VOC analysis woth electronic nose and mass spectrometry. VOC profiles will be compared between the two groups of patients.

DETAILED DESCRIPTION:
Prospective single-center study. A single visit, no follow-up. The visit will take place before or within five days from date of transbronchial biopsies (BTB). It will include a noninvasive collection of exhaled breath for VOC analysis. VOC analysis will be conducted using two types of devices: "electronic nose" and mass spectrometry.

200 bi-lung transplanted patients will be enrolled and divided into two groups.

* Group A, Acute rejection: 100 patients. Diagnosis of acute rejection retained on transbronchial biopsies or functional anomalies with the necessity of modifying the immunosuppressive regimen.
* Group B, control: 100 patients. Patients without respiratory functional abnormality and normal transbronchial biopsy.

VOC, detected by electronic nose and identified by mass spectrometry, will be compared between patients with a confirmed diagnosis of acute rejection (group A) and patients without rejection (control group B)

The duration of participation of each patient is 1 day. The duration of the inclusion period is estimated at 54 months from the first inclusion. The expected total duration of the research is 54 months

ELIGIBILITY:
Inclusion Criteria:

* Bi-pulmonary transplant patient
* Acute rejection group: Patients with transbronchial biopsies performed as part of their usual follow-up or for functional abnormality ; Diagnosis of acute rejection retained on the following arguments: histological lesions of cellular rejection or histological lesions of humoral rejection or normal histology but diagnosis of "functional rejection" retained and immunosuppressive treatment indicated
* Control group: Patients benefiting from systematically programmed transbronchial biopsies as part of post-transplant follow-up with normal histology and absence of functional respiratory abnormality

Exclusion Criteria:

* Patient unable to realize a vital capacity measure
* Neoplasia currently treated
* Unresolved acute bronchial complication (stenosis or dehiscence)
* Immunosuppressive treatment of acute rejection already begun
* Patient who has already participated in the protocol and already included in one of the two study groups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-06-27 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Volatile Organic Compounds by electronic nose (eNose) | 1 day
  Comparison of Volatile Organic Compounds profile detected by electronic nose between lung transplant patients patients with a confirmed diagnosis of acute rejection and patients without rejection

SECONDARY OUTCOMES:
Volatile Organic Compounds profile | 1 day
  Comparison of Volatile Organic Compounds profile identified by mass spectrometry electronic nose between lung transplant patients with a confirmed diagnosis of acute rejection and patients without rejection
Acute rejection diagnosis | 1 day
  Comparison of discriminative capacity for diagnosis of acute rejection between the VOC analysis methods: electronic nose versus mass spectrometry.
Volatile Organic Compounds by spectrometry | 1 day
  Determining distinct exhaled VOC profiles associated with each type of acute rejection: cellular rejection, humoral rejection or functional rejection

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Couderc, MD-PhD, Study Chair — Pneumologie Hopital Foch; Antoine Roux, Principal Investigator — Pneumologie Hopital Foch; Hélène Salvator, MD, Study Chair — Pneumologie Hopital Foch; Philippe Devillier, MD-PhD, Study Chair — UPRES EA 220 Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No